CLINICAL TRIAL: NCT04833426
Title: Impact of Peri-operative tEstosterone Levels on oNcological and Functional Outcomes in RadiCal prostatEctomy
Acronym: ENFORCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canisius-Wilhelmina Hospital (Other)
Collaborators: Besins Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL7436209120; 2020-003012-27 (EudraCT Number); 2020-6874 (Other: CMO Arnhem-Nijmegen)
Record Dates: First submitted 2021-02-05; First posted 2021-04-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms; Hypogonadism; Testosterone Deficiency
Keywords: Prostate cancer; Prostatectomy; Hypogonadism; Testosterone deficiency
MeSH Terms: conditions — Prostatic Neoplasms; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone therapy (Active Comparator): Daily application of two pump auctions of 16.2mg/ml testosterone gel. Dosage may be altered depending on clinical response
  Interventions: Drug: Testosterone gel
- Placebo therapy (Placebo Comparator): Daily application of two pump auctions of placebo gel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone gel — Topical gel containing testosterone
  Other Names: Androgel
  Arms: Testosterone therapy
Drug: Placebo — Topical gel without active substance
  Other Names: Placebo gel
  Arms: Placebo therapy

SUMMARY:
Sexual dysfunction is a common side effect of radical prostatectomy (RP) and has a significant negative impact on quality of life. With age the testosterone level in men declines; around 30% of men over 70 years of age meet the criteria of testosterone deficiency (TD). The negative impact of both TD and RP on sexual performance are likely to add up. The aim of this study is to assess the efficacy and safety of testosterone replacement therapy (TRT) on functional and oncological outcomes in testosterone deficient men following RP for prostate cancer (PCa).

DETAILED DESCRIPTION:
Rationale: Radical prostatectomy (RP) is currently the most common treatment for non-metastatic prostate cancer (PCa). Two frequent side effects of this procedure are urinary incontinence and erectile dysfunction, both having a significant negative impact on quality of life.

Additionally, it is known that with age the testosterone level in men declines. This does not lead to symptoms in all men (asymptomatic testosterone deficiency). Both testosterone deficiency (TD) and radical prostatectomy are well-established to have a significant negative impact on sexual performance and are likely to add up in patients with a low testosterone following RP.

Objective: The aim of this study is to assess the effect of testosterone replacement therapy (TRT) on functional and oncological outcomes in testosterone deficient men following RP for PCa.

Study design: This study is a phase 3 prospective, randomized, placebo-controlled, single-blind clinical trial. Study population: All men over 18 years old diagnosed with non-metastatic prostate cancer who are scheduled for RP within three months as primary treatment, can be prescreened for inclusion. Prior to the RP, serum testosterone will be determined. Subsequently, within six weeks after the RP, serum testosterone will be determined again and patients will be screened for inclusion. If necessary, a third measurement of testosterone will be done. Eligible patients meet the criteria for TD and other inclusion criteria. Intervention: Patients will be randomized for testosterone replacement therapy (TRT) or placebo as a daily administered topical gel starting within 8 weeks after RP. Patients will receive TRT or placebo for one year following RP and will be monitored for another year for functional outcomes and for four more years to establish 5-year biochemical recurrence (BCR) free survival.

Main study parameters/endpoints:

The primary study endpoint is a clinically relevant (12 points or more) difference in the EPIC-26 domain for sexual functioning 12 months after RP in favor of testosterone deficient men receiving TRT compared with testosterone deficient men receiving placebo. Secondary endpoints include: urinary incontinence score, hormonal functioning score and BCR-free survival. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The number of visits and blood drawings are equal to standard of care follow-up after RP, with the exception of two or three extra blood samples at the first prescreening visit and within six weeks following RP. We ask patients to remain with their hospital for 24 months after RP for follow-up and to complete online questionnaires for the given visits. The five-year biochemical recurrence (BCR) free survival will be obtained through patient's medical records and if insufficient, through the Dutch Cancer Registry (NKR). Patients who receive TRT or placebo can experience local side-effects such as itching, rash and/or irritation at the site of application. In addition, patients who receive TRT can experience systemic sideeffects are gain of weight, hot flashes, acne and an increase in red blood count level. Furthermore, TRT might improve sexual functioning, urinary continence, hormonal functioning and BCR-free survival, but this is not certain and is subject of research in this study.

ELIGIBILITY:
Inclusion criteria

1. Men aged 18 years or older
2. Histologically confirmed prostate cancer
3. Radical prostatectomy performed as primary treatment
4. At least one-sided nerve-sparing procedure performed
5. Non-metastatic disease (cN0M0) based on the use of nomograms or imaging
6. Undetectable PSA level (<0.1 µg/l or unmeasurable according to local protocol) within six weeks following RP
7. A preoperative minimal sexual function, defined as a score of 40 points or more (out of 100) for the EPIC-26 sexual function domain
8. Testosterone deficiency, defined as total testosterone <8 nmol/L, or total testosterone between 8-12 nmol/L with free testosterone <225 pmol/L, measured on two separate occasions, with normal or elevated luteinising hormone (LH)

Exclusion criteria

1. Prior prostate cancer treatment, including but not limited to anti-hormonal therapy, radiotherapy, or brachytherapy (active surveillance allowed)
2. Previous use of testosterone therapy for any reason
3. Pathological stage pT3b or pT4 in the RP specimen
4. Positive surgical margin(s) with ISUP grade 4 or 5 in the RP specimen
5. Presence of metastatic lymph nodes if pelvic lymph node dissection was performed
6. History of male breast cancer or liver tumour
7. Uncontrolled hypertension
8. General contraindications for TRT
9. Allergy for components in TRT agent or placebo
10. Use of vitamin K antagonists
11. Body mass index (BMI) >30 kg/m²

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant (≥12 points) difference in the EPIC-26 sexual functioning domain score, 12 months after radical prostatectomy between groups. | 12 months
  Functional recovery after radical prostatectomy will be assessed by EPIC-26 questionnaire, a Patient Reported Outcome Measure (PROM). Patients will be asked to complete this questionnaire online.

SECONDARY OUTCOMES:
Clinically relevant (≥12 points) difference in the EPIC-26 sexual functioning domain score 3 months after radical prostatectomy between groups. | 3 months
  Clinical relevance (>12 points) for sexual function domain score as measured by EPIC-26.
Clinically relevant (≥12 points) difference in the EPIC-26 sexual functioning domain score 24 months after radical prostatectomy between groups. | 24 months
  Clinical relevance (>12 points) for sexual function domain score as measured by EPIC-26.
Clinically relevant (≥9 points) difference in the EPIC-26 urinary incontinence domain score, 12 months after radical prostatectomy between groups. | 12 months
  Clinical relevance (>9 points) for Urinary incontinence domain score as measured by EPIC-26.
Clinically relevant (≥9 points) difference in the EPIC-26 urinary incontinence domain score, 24 months after radical prostatectomy between groups. | 24 months
  Clinical relevance (>9 points) for Urinary incontinence domain score as measured by EPIC-26.
Clinically relevant (≥6 points) difference in the EPIC-26 for hormonal functioning domain score, 12 months after radical prostatectomy between groups. | 12 months
  Clinical relevance (>6 points) for hormonal functioning domain score as measured by EPIC-26.
Clinically relevant (≥6 points) difference in the EPIC-26 for hormonal functioning domain score, 24 months after radical prostatectomy between groups. | 24 months
  Clinical relevance (>6 points) for hormonal functioning domain score as measured by EPIC-26.
Difference in biochemical recurrence rate between groups. | 5 years
  Biochemical recurrence (BCR) is defined as the occurrence of measurable (>0.1 ng/ml) prostate specific antigen (PSA), during routinely follow-up up to five years after surgery, determined at two different occasions with at least one week between them.The BCR-rate between the placebo and control group will be compared to determine the influence of testosterone therapy on BCR.

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Somford, MD, PhD, Principal Investigator — Canisius-Wilhelmina Hospital
Locations (10):
- Netherlands (10):
  - Amsterdam UMC location VUmc, Amsterdam
  - Netherlands Cancer Institute, Amsterdam
  - Rijnstate, Arnhem
  - Catharina Hospital, Eindhoven
  - Treant, Emmen
  - Zuyderland, Heerlen
  - St. Antonius Hospital, Nieuwegein
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud university medical center, Nijmegen
  - Máxima Medical Centre, Veldhoven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baas D, van Drumpt J, Kiemeney L, Beck J, Ostergren PB, Sedelaar M, Hoekstra R, Spruyt AB, van Melick H, Bruins M, van Leeuwen P, Vis A, Wijburg C, Roelofs L, van den Bergh R, van Soest R, van Basten JP, Somford D. Clinical Trial Protocol: Impact of Testosterone Replacement Therapy on Functional and Oncological Outcomes Following Radical Prostatectomy (ENFORCE Study). Eur Urol Oncol. 2025 Jun 12:S2588-9311(25)00168-3. doi: 10.1016/j.euo.2025.05.024. Online ahead of print. PMID 40514343

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT04833426/Prot_SAP_000.pdf